CLINICAL TRIAL: NCT05765565
Title: Comparison Between the Multi-electrode Octaray and Pentaray Catheters in Patients Undergoing Ablation for Atrial Tachycardia Using Coherent Mapping.
Brief Title: Comparison Between the Octaray and Pentaray Catheters in Patients Undergoing Ablation for Atrial Tachycardia.
Acronym: OCTOPUS-AT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Tamas Szili-Torok, Dr., Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC-2022-0269
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Atrial Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octaray (intervention) (Experimental): Octaray created 3D map quality
  Interventions: Device: Octaray multi-electrode catheter
- Pentaray (control) (Active Comparator): Pentaray created 3D map quality
  Interventions: Device: Pentaray multi-electrode catheter

INTERVENTIONS:
Device: Octaray multi-electrode catheter — Newly designed multi-electrode catheter for creating 3D electroanatomical CARTO maps.
  Arms: Octaray (intervention)
Device: Pentaray multi-electrode catheter — Current standard multi-electrode catheter for creating 3D electroanatomical CARTO maps.
  Arms: Pentaray (control)

SUMMARY:
The goal of this randomized clinical trial is to compare the 3D electroanatomical activation map-quality and -efficiency in patients undergoing atrial tachycardia (AT) catheter ablation. Primary objective of the study is to contrast CARTO-Coherent mapping quality (electrograms per map) using Octaray versus Pentaray catheter for left and right atrium ATs, separately.

Participants will be randomized with 1:1 ratio for undergoing 3D anatomy map with either Octaray (intervention group) or Pentaray (control) group. Next, all patients will undergo activation map of the AT with both catheters. For ablation in the intervention group, the Ocatray made activation map of the AT will be used, and the Pentary made AT activation map will be used in the control group.

DETAILED DESCRIPTION:
This is a randomized open-label cross-over trial including consecutive patients undergoing ablation for atrial tachycardia of the left and right atrium. The sample-sizes of the left (N=20) and right (N=20) atrium will be equal. Half of the eligible patients with either left or right atrium AT will be randomized to undergo Coherent Mapping with Pentaray catheter first followed by Coherent Mapping with the Octaray catheter. The other half will undergo initial Coherent Mapping with the Octaray catheter followed by Pentaray catheter. This way all study participants (total N=40) will undergo the Coherent Mapping with both catheters (Figure 1). Only the second map created with either Octaray (n active arm left atrium =10 and n active arm right atrium =10) or Pentaray (n control arm left atrium =10 and n control arm right atrium =10) will be used for the subsequent ablation procedure.

The main outcome of the trial is the performance of the Coherent Mapping quality (electrograms per map) with Octaray catheter versus Pentaray catheter for left and right atrium, separately. A map will be considered complete when the fill threshold reach 5 mm for the entire surface area of the left or right atrium, that is the interpolation between points will be <5 mm as previously reported. The high- and low-pass filters settings will be harmonized between the catheters. The following data will be collected: 1) number of electrograms per map; 2) Voltage based signal-to-noise ratio (vSNR),17 calculated as the ratio between the mean of the peak-to-peak amplitude of the true local bipolar atrial signals and the mean of the SD of the peak-to-peak of all other signals considered as far-field or ambient lab noise; 3) electrograms acquisition rate (i.e., the acquired number of points per minute of mapping); 4) electrograms acquisition density (i.e., the acquired number of electrograms per cm2 of the left or right atrium); 5) number of electrograms acquired per beat; 6) the total ablation and fluoroscopy times; 7) acute mapping success rate, defined as termination of AT at the target region; 8) number of entrainments attempted and the best post-pacing interval value at the ablation site when available. Successful entrainment is sometimes not possible (i.e., focal AT) and some investigator may prefer not to entrain. Therefore, the decision to use entrainment and the number of entrainment attempts will be left to the discretion of the operator.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Planned for catheter ablation of either left- or right-atrium AT/flutter will be eligible for inclusion. In the group of right atrium AT patients with typical flutters will also be eligible for inclusion.

Exclusion Criteria:

* Individuals not able to provide informed consent for any reason including language and mental disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-21 (Estimated); Primary Completion 2024-03-21 (Estimated); Study Completion 2024-03-21 (Estimated)

PRIMARY OUTCOMES:
Number of electrograms per map | during procedure

SECONDARY OUTCOMES:
Voltage based signal-to-noise ratio. | during procedure
electrograms acquisition rate | during procedure
  the acquired number of points per minute of mapping)
electrogram acquisition density | during procedure
  the acquired number of electrograms per cm2 of the left or right atrium
number of electrograms acquired per beat | during procedure
the total ablation and fluoroscopy times | during procedure
acute mapping success rate | during procedure
  defined as termination of AT at the target region
number of entrainments attempted and the best post-pacing interval value at the ablation site | during procedure
  May not be available especially in focal AT's

IPD SHARING:
Plan to Share IPD: Undecided
Needs to be discussed with the catheter manufacturer